CLINICAL TRIAL: NCT03449121
Title: Pilot Study for Breathing Interventions in Congestive Heart Failure
Brief Title: Study for Breathing Interventions in Congestive Heart Failure
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left VUMC
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 171991
Record Dates: First submitted 2018-01-31; First posted 2018-02-28 (Actual); Last update posted 2019-03-04 (Actual); Status verified 2019-02

CONDITIONS: Congestive Heart Failure
Keywords: Breathing; Mind-body
MeSH Terms: conditions — Heart Failure; Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Slow breathing (Experimental): Slow breathing techniques with exhale greater than inhale
  Interventions: Behavioral: Slow breathing techniques

INTERVENTIONS:
Behavioral: Slow breathing techniques — 8 sessions of instruction in slow breathing exercises over 12 weeks of study

SUMMARY:
Slow breathing may reduce stress. Adults with congestive heart failure have higher stress than the general population. This study will examine if using slow breathing is feasible among adults with heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Documented heart failure from medical chart review with signs and symptoms consistent with disease
* Reduced left ventricular function with ejection fraction of less than or equal to 40%
* English speaking

Exclusion Criteria:

* New York Heart Failure Association Class I or IV
* Myocardial infarction in the last 3 months
* Cardiac surgery in the last 3 months
* Significant valvular heart disease
* Uncontrolled cardiac arrhythmias
* Uncontrolled diabetes mellitus (hemoglobin a1c ≥ 8)
* Uncontrolled hypertension
* Systolic greater than 140 mmHg
* Diastolic greater than or 90 mmHg
* Cognitive impairment (Mini-mental state exam less than or equal to 24)
* Acute major depression in the last 3 months
* Other psychiatric conditions including schizophrenia or bipolar disorder
* Attention-deficit-disorder or attention-deficit-hyperactivity disorder
* Musculoskeletal condition limiting capacity to perform simple movements such as significant chronic lower back pain or neck pain
* Unstable or severe chronic lung conditions
* Current participation in a mind-body practice/program
* Current cancer other than non-melanoma skin cancer
* Regular swimmer
* Plays wind or brass musical instruments

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-11 (Estimated); Primary Completion 2019-05 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Feasibility of intervention administration measured by frequency of visits | Weekly for 12 weeks
  Investigators will document weekly attendance
Feasibility of intervention administration measured by home practice adherence | Weekly for 12 weeks
  Investigators will ask participants how often they practiced yoga at home since last session
Feasibility of intervention administration measured by patient satisfaction | One time, at 12 week survey
  A survey will be administered that assesses participant satisfaction with the yoga. Overall satisfaction will be assessed by "Very Unsatisfied", "Unsatisfied", "Satisfied", "Very Satisfied".
Safety of yoga practice as measured by occurrence of adverse events | Weekly for 12 weeks
  Investigators will monitor for adverse events related to yoga practice during the intervention and will solicit any adverse events during home practice since last meeting.

SECONDARY OUTCOMES:
Magnitude of change in PROMIS Depression scale | Baseline, 6 week, 12 week
  Patient-Reported Outcomes Measurement Information System (PROMIS) Depression Computer Adaptive Test (CAT). The PROMIS Depression instruments assess self-reported negative mood (sadness, guilt), views of self (selfcriticism, worthlessness), and social cognition (loneliness, interpersonal alienation), as well as decreased positive affect and engagement (loss of interest, meaning, and purpose). With CAT, participant responses guide the system's choice of subsequent items from the full item bank (28 items in total) and a T-Score is generated. T-Score distributions are standardized such that a 50 represents the average (mean) for the US general population, and the standard deviation around that mean is 10 points. A higher score reflects higher levels of depression.
Magnitude of change in PROMIS Anxiety scale | Baseline, 6 week, 12 week
  Patient-Reported Outcomes Measurement Information System (PROMIS) Anxiety Computer Adaptive Test (CAT). The PROMIS Anxiety instruments measure self-reported fear (fearfulness, panic), anxious misery (worry, dread), hyperarousal (tension, nervousness, restlessness), and somatic symptoms related to arousal (racing heart, dizziness). With CAT, participant responses guide the system's choice of subsequent items from the full item bank (29 items in total) and a T-Score is generated. T-Score distributions are standardized such that a 50 represents the average (mean) for the US general population, and the standard deviation around that mean is 10 points. A higher score reflects higher levels of anxiety.
Magnitude of change in PROMIS Global Health scale | Baseline, 6 week, 12 week
  Patient-Reported Outcomes Measurement Information System (PROMIS) Global Health. The PROMIS Global Health measures assess an individual's physical, mental, and social health. Each of the 10 items are totaled into a raw sum score and Raw Sum Scores are then converted into T-Scores. T-Score distributions are standardized such that a 50 represents the average (mean) for the US general population, and the standard deviation around that mean is 10 points. A higher score reflects higher levels of physical, mental, and social health.
Magnitude of change in PROMIS Physical Function scale | Baseline, 6 week, 12 week
  Patient-Reported Outcomes Measurement Information System (PROMIS) Physical Function Computer Adaptive Test (CAT). PROMIS Physical Function instruments measure self-reported capability rather than actual performance of physical activities. This includes the functioning of one's upper extremities (dexterity), lower extremities (walking or mobility), and central regions (neck, back), as well as instrumental activities of daily living, such as running errands. With CAT, participant responses guide the system's choice of subsequent items from the full item bank (165 items in total) and a T-Score is generated. T-Score distributions are standardized such that a 50 represents the average (mean) for the US general population, and the standard deviation around that mean is 10 points. A higher score reflects higher levels of physical functioning.
Magnitude of change in PROMIS Fatigue scale | Baseline, 6 week, 12 week
  Patient-Reported Outcomes Measurement Information System (PROMIS) Fatigue Computer Adaptive Test (CAT). The PROMIS Fatigue instruments evaluate a range of self-reported symptoms, from mild subjective feelings of tiredness to an overwhelming, debilitating, and sustained sense of exhaustion that likely decreases one's ability to execute daily activities and function normally in family or social roles. With CAT, participant responses guide the system's choice of subsequent items from the full item bank (95 items in total) and a T-Score is generated. T-Score distributions are standardized such that a 50 represents the average (mean) for the US general population, and the standard deviation around that mean is 10 points. A higher score reflects higher levels of fatigue.
Magnitude of change in PROMIS Dyspnea scale | Baseline, 6 week, 12 week
  Patient-Reported Outcomes Measurement Information System (PROMIS) Dyspnea Severity Computer Adaptive Test (CAT). The PROMIS Dyspnea instruments evaluate a range of self-reported symptoms related to dyspnea. With CAT, participant responses guide the system's choice of subsequent items from the full item bank (33 items in total) and a T-Score is generated. T-Score distributions are standardized such that a 50 represents the average (mean) for the US general population, and the standard deviation around that mean is 10 points. A higher score reflects higher levels of dyspnea.
Autonomic tone | Monthly data extraction from ICD: Baseline, week 4, week 8, week 12
  The investigators will estimate autonomic tone of participants by extracting data from implantable cardioverter defibrillator (ICD). Data analyses will consist of heart rate spectral analyses.

IPD SHARING:
Plan to Share IPD: No